CLINICAL TRIAL: NCT01488552
Title: A Phase II Study of Induction Consolidation and Maintenance Approach for Patients With Advanced Pancreatic Cancer
Brief Title: Gemcitabine+Nab-paclitaxel and FOLFIRINOX and Molecular Profiling for Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pancreatic Cancer Research Team (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCRT 11-002
Record Dates: First submitted 2011-11-18; First posted 2011-12-08 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Stage IV Pancreatic Cancer
Keywords: pancreatic cancer; pancreatic adenocarcinoma; Stage IV pancreatic cancer; pancreas; pancreatic
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; folfirinox; Fluorouracil; Immunohistochemistry; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine & Abraxane Pancreatic Cancer (Experimental): Gemcitabine+Nab-paclitaxel, FOLFIRINOX, Immunohistochemistry (IHC) Analysis, Metformin and Folfiri
  Interventions: Drug: Gemcitabine; Drug: nab-paclitaxel; Drug: FOLFIRINOX; Genetic: Immunohistochemistry (IHC) Analysis; Drug: Metformin; Drug: mFOLFIRI

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m2 weekly on days 1,8, and 15 in a 28 day cycle. Part A: nab-paclitaxel/Gem for 6 cycles, followed by FOLFIRINOX for 6 cycles (31 patients); Part B: Alternate nab-paclitaxel/Gem with mFOLFIRI every 2 months for up to 1 year or 6 cycles of each regimen (30 patients).
  Other Names: Gemzar
Drug: nab-paclitaxel — 125 mg/m2 on days 1,8, and 15 of a 28 day cycle Part A: nab-paclitaxel/Gem for 6 cycles, followed by FOLFIRINOX for 6 cycles (31 patients); Part B: Alternate nab-paclitaxel/Gem with mFOLFIRI every 2 months for up to 1 year or 6 cycles of each regimen (30 patients).
  Other Names: Abraxane
Drug: FOLFIRINOX — The combination below will be given on days 1 and 15 of a 28 day cycle; 5-Fluorouracil 2400 mg/m2 with a 46-hour continuous IV infusion; Leucovorin 400 mg/m2 over a 2 hour IV infusion;
  Oxaliplatin 85 mg/m2 as a 2 hour IV infusion; Irinotecan 180 mg/m2 over a 90 minute IV infusion Part A: nab-paclitaxel/Gem for 6 cycles, followed by FOLFIRINOX for 6 cycles (31 patients); Part B: Alternate nab-paclitaxel/Gem with mFOLFIRI every 2 months for up to 1 year or 6 cycles of each regimen (30 patients).
  Other Names: 5-FU; Eloxitan; Campostar
Genetic: Immunohistochemistry (IHC) Analysis — Immunohistochemistry (IHC) Analysis will be performed on a fresh tissue biopsy of the tumor after chemotherapy has been administered. A targeted-based regimen will be determined from the results of the IHC analysis for the next therapy given to the patient in the maintenance phase of the study.
Drug: Metformin — Metformin 500 mg daily as a 24 hour extended release tablet will also be given as part of the maintenance phase of this study.
  Other Names: Glucophage
Drug: mFOLFIRI — 5-FU IV infusion, 2400 mg/m2 46h continuous infusion (no bolus 5-FU) treatments per month equaling 1 cycle Leucovorin 400 mg/m2 dl (over a 2 hour IV infusion) Irinotecan 180 mg/m2 dl (over a 90 minute IV infusion) Part A: nab-paclitaxel/Gem for 6 cycles, followed by FOLFIRINOX for 6 cycles (31 patients); Part B: Alternate nab-paclitaxel/Gem with mFOLFIRI every 2 months for up to 1 year or 6 cycles of each regimen (30 patients).

SUMMARY:
The Investigators in the PCRT team have developed a therapeutic regimen which attacks both the tumor compartment and the stromal compartment of pancreatic cancer and induces complete responses in a small percentage of patients with advanced stage IV pancreatic cancer.

DETAILED DESCRIPTION:
The investigators in the PCRT team have developed a therapeutic regimen which attacks both the tumor compartment and the stromal compartment of pancreatic cancer and induces complete responses in a small percentage of patients with advanced stage IV pancreatic cancer.

The gemcitabine + nab-paclitaxel regimen had outstanding activity in a 67 patient phase I/II trial with all patients at the recommended phase II doses (n=44) having a decrease in CA19-9, some complete responses and a median survival of 12.2 months. The proposed regimen that is devised for this study is a bold, innovative approach with the specific aim of utilizing a relentless pursuit approach to try to make the complete response rate >70% and have this response be durable (which the PCRT has defined as lasting at least 6 months) and to dramatically enhance the percent of patients who survive one year (try to make the rate >70%).

The induction regimen the investigators propose collapses the stroma (gemcitabine + nab-paclitaxel) and addresses the use of a non-cross resistant active regimen (FOLFIRINOX) as a consolidation regimen. Both should improve the chance of driving tumor markers down dramatically. The investigators think that FOLFIRINOX with the stromal collapse induced by the initial regimen, plus the totally non-cross resistant shot against the disease (consolidation), will maximize the chance of achieving a complete response with an attendant improvement in survival.

After the consolidation, the patient will be maintained on a less toxic targeted therapy selected by molecular profiling plus the use of the antimetabolomic agent metformin which has consistently been associated with better survival in multiple retrospective studies (Jiralerspong et al., 2009).

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented Stage IV metastatic adenocarcinoma of the pancreas with measurable disease
* Performance status ECOG 0 or 1
* Patients may not have received prior treatment for metastatic pancreatic adenocarcinoma except for receiving gemcitabine or 5FU as a radiosensitizer along with radiation therapy; or have received gemcitabine for adjuvant treatment if they have been off gemcitabine for > 12 months
* Adult (>18 years of age) male or non-pregnant and non-lactating female
* A negative serum pregnancy test (Beta-hCG) documented within 72 hours of the first administration of study drug in female patients of child-bearing potential
* Agreement to use contraception considered adequate and appropriate by the investigator
* The following blood counts at baseline:

  * ANC >/= 1.5 x 109/L
  * Hgb > 9g/dL
  * Platelets >100 x 109/L
* The following blood chemistry levels at baseline:

  * AST and ALT </= 2.5 x upper limit of normal range (ULN) or < 5.0 ULN if liver metastasis are present
  * Bilirubin </= ULN
  * Serum creatinine within 1.5 x ULN
* PT, INR within 1.5 x ULN unless on therapeutic doses of warfarin
* Must have measurable disease outside the pancreas by RECIST criteria
* No clinically significant abnormalities in urinalysis results
* Voluntary agreement to participate in this study after being informed about the nature of the study including potential risks and benefits and having the ability to have questions addressed. The patient must sign and date the IRB approved Informed Consent Form (ICF) prior to participation in any study-related procedures

Exclusion Criteria:

* Has pancreatic islet cell neoplasms
* Is pregnant or lactating
* Has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* Known infection with HIV, Hepatitis B or Hepatitis C.
* Patient with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies (see section 4.4.9)
* Has a serious medical risk factor(s) involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive an experimental research drug.
* Is unwilling or unable to comply with study procedures.
* Is enrolled in any other investigational trial.

Caution of observation for interstitial pneumonitis in patients prior to enrollment:

Before enrollment, evaluate candidate patients fro familial, environmental or occupational exposure to opportunistic pathogens, and do not enroll those with a history of slowly progressive dyspnea and unproductive cough, or of conditions such as sarcoidosis, silicosis. idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Complete Response Rate | 1 yr.
  The primary objectives of this study are to relentlessly pursue treatment for 34 individual patients with Stage IV pancreatic cancer to obtain:
  • The complete response rate (as defined by a complete metabolomic response (CMR) of SUV normalization from baseline, OR a complete response on CT scan using a modified RECIST criteria and CA 19-9 (or CA 125, CEA, or PAM4 if not expressers of CA 19-9) down to normal limits (from at least > 2X ULN).

SECONDARY OUTCOMES:
One-Year Survival Endpoint | 1 yr.
  A secondary objective of this study is to:
  Observe the percent of patients who are alive at one year (our goal is to obtain a >70% one year survival.)
Efficacy Endpoints using biomarkers | 1 yr.
  A secondary objective of this study is to:
  Gather information on other possible efficacy endpoints (e.g. CA 19-9) and other serum/plasma tumor markers
Observing toxicity outcomes | 1 yr.
  A secondary objective of this study is to document the toxicities noted in all patients, particularly with those who receive the FOLFIRINOX regimen. Grade 3-4 neutropenia is expected to be > 40% among those receiving FOLFIRINOX, so to minimize toxicity, all patients will receive prophylactic CGSF. In the first 9 patients receiving FOLFIRINOX, if the hospitalization rate due to toxicity is more than 50% (5 or more patients), then all subjects will have a dose reduction to level -1. The incidence of grade 3 and 4 toxicities and dose delays will also be considered for dose modification.

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh K Ramanathan, MD, Principal Investigator — Translational Genomics Research Institute
Locations (5):
- United States (5):
  - TGen Clinical Research Services (TCRS), Scottsdale, Arizona
  - Disney Family Cancer Center, Burbank, California
  - Virginia Piper Cancer Institute (VPCI), Minneapolis, Minnesota
  - Virginia Mason Medical Center, Seattle, Washington
  - Evergreen Hematology and Oncology, Spokane, Washington

REFERENCES:
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Von Hoff DD, Ramanathan RK, Borad MJ, Laheru DA, Smith LS, Wood TE, Korn RL, Desai N, Trieu V, Iglesias JL, Zhang H, Soon-Shiong P, Shi T, Rajeshkumar NV, Maitra A, Hidalgo M. Gemcitabine plus nab-paclitaxel is an active regimen in patients with advanced pancreatic cancer: a phase I/II trial. J Clin Oncol. 2011 Dec 1;29(34):4548-54. doi: 10.1200/JCO.2011.36.5742. Epub 2011 Oct 3. PMID 21969517
- See also: Additional information about the Pancreatic Cancer Research Team (PCRT) — http://www.pcrt.org
- See also: Non-profit Organization — http://www.tgen.org
- See also: Related link — http://www.td2inc.com
- See also: Non-profit organization for pancreatic cancer research — http://www.seenamagowitzfoundation.org/